CLINICAL TRIAL: NCT00401739
Title: Phase I Study of CSL360 in Patients With Relapsed, Refractory or High-Risk Acute Myeloid Leukemia
Brief Title: Safety, Tolerability and Pharmacokinetics of CSL360 in the Treatment of Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Limited (Industry)
Responsible Party: Dr Russell Basser, CSL Limited
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-AML-06-26
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CSL360

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Treatment with CSL360
  Interventions: Drug: CSL360

INTERVENTIONS:
Drug: CSL360 — Weekly IV Infusion. Dose escalation study.

SUMMARY:
Acute myeloid leukemia (AML) is a heterogeneous group of diseases characterized by uncontrolled proliferation of the myeloid line of white blood cells and impaired production of normal blood cells. If untreated, patients die of infection or bleeding usually in a matter of weeks. CSL360 is a neutralising monoclonal antibody which is believed to target the cells that are thought to drive AML but that are not effectively killed by standard treatment. The aims of the study are to determine a biologically active dose of CSL360 and generate understanding of a rational schedule of administration for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute myeloid leukemia
* Recent bone marrow biopsy
* Prior treatment or medically unfit for standard therapy

Exclusion Criteria:

* Peripheral blood blast count > 30 x 109/L, or rapidly progressive AML
* Previous solid organ transplant
* Active GvHD or immunosuppression
* Concurrent treatment with other anti-cancer therapy
* Active infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Adverse events, pharmacokinetics | September 2009

SECONDARY OUTCOMES:
Maximum tolerated dose | September 2009
Partial, complete and overall response | September 2009
Biological activity | September 2009

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Roberts, Dr, Principal Investigator — Melbourne Health
Locations (6):
- Australia (6):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Institute of Medical & Veterinary Science, Adelaide, South Australia
  - Peter MacCallum Cancer Institute, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria